CLINICAL TRIAL: NCT03659383
Title: The Exploration of Optimal Treatment Scheme in Patients With Type 2 Diabetes Inadequately Controlled With Glargine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20170904-03
Record Dates: First submitted 2018-06-12; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-06

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Optimal hypoglycemic treatment (Experimental): The patients will receive optimal hypoglycemic treatments, including adjustment of insulin dose and oral antidiabetic agents
  Interventions: Combination Product: Optimal hypoglycemic treatment

INTERVENTIONS:
Combination Product: Optimal hypoglycemic treatment — Standardize oral hypoglycemic medication and adjust insulin dose according to blood glucose values obtained by self-monitoring

SUMMARY:
Glargine is commonly used in insulin supplemental therapy in patients with type 2 diabetes(T2D) at present. However, many patients who treated with glargine still have poor blood glucose control because of insufficient insulin dose or improper oral medication. This study aims to investigate the optimal treatment scheme in order to improve the blood control in these patients. Continuous Glucose Monitoring System (CGMS) will be used to assess the blood glucose control at baseline and the moment when the patients achieved standard. Oral medications will be standardized first, and insulin doses will be adjusted according to blood glucose values obtained by self-monitoring. Glycemic control will be considered as reaching target of glucose if the fasting capillary blood glucose is less than 6.1 mmol/L. The maximum period of blood glucose adjustment will be 1 months. Oral medication, the type and dosage of insulin, exercise status, insulin injection skill evaluation, islet function, duration of diabetes, complications and insulin antibodies will be recorded in detail at baseline, reaching target of glucose standard and 3 months after reaching target of glucose.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with T2DM, which was defined bypublished Criteria of World Health Organization in 1999;
2. Patients were using glargine with or without oral hypoglycemic drugs and having a stable dose of glargine for more than 2 month would be recruited into this study;
3. Patients had relatively constant diet and exercise in 2 month before the study.
4. Fasting blood glucose was between 6.1 and 16mmolL, and postprandial (or random) blood glucose <22.2mmol/L

Exclusion Criteria:

1. Patients with severe cardiovascular diseases, such as stroke, transient ischemic attack, myocardial infarction, unstable angina, coronary artery bypass grafting, percutaneous coronary intervention, and heart failure;
2. Patients with severe infectious diseases;
3. Patients with acute complications of diabetes on admission, such as diabetic ketoacidosis, diabetic hyperosmolar nonketotic coma, and lactic acidosis;
4. Patients with history of psychiatric disorders and were unsuitable to use CGMS;
5. Any other situations that made patients unsuitable to participate in the study, such as alcoholism and drug abuse.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-09-20 (Estimated); Primary Completion 2019-02-20 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Rate of reaching target of glucose | 0-1 month
  Rate of reaching target of glucose

SECONDARY OUTCOMES:
HbA1c | 0-3 month
  Glycated hemoglobin at baseline and 3 months after reaching target of blood glucose
Dosage of insulin | 0-1 month
  Change of insulin dose
Time of reaching target of glucose | 0-1 month
  Time of reaching target of glucose